CLINICAL TRIAL: NCT06600321
Title: A Phase 1 Study of ALN-BCAT as Monotherapy and in Combination With Pembrolizumab in Patients With Advanced or Metastatic Hepatocellular Carcinoma
Brief Title: A Study to Evaluate ALN-BCAT in Patients With Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALN-BCAT-001
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Advanced Hepatocellular Carcinoma; Metastatic Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma (HCC); Pembrolizumab; CTNNB1; Liver disease; Liver cancer; Liver neoplasms; Carcinoma, hepatocellular; WNT pathway activating
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Diseases; Liver Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Monotherapy: Dose Escalation (Experimental): Patients will be administered multiple doses of ALN-BCAT.
  Interventions: Drug: ALN-BCAT
- Monotherapy: Dose Expansion (Experimental): Patients will be administered multiple doses of ALN-BCAT.
  Interventions: Drug: ALN-BCAT
- Combination Therapy: Dose Escalation (Experimental): Patients will be administered multiple doses of ALN-BCAT in combination with pembrolizumab.
  Interventions: Drug: ALN-BCAT; Drug: Pembrolizumab
- Combination Therapy: Dose Expansion (Experimental): Patients will be administered multiple doses of ALN-BCAT in combination with pembrolizumab.
  Interventions: Drug: ALN-BCAT; Drug: Pembrolizumab

INTERVENTIONS:
Drug: ALN-BCAT — Administered by intravenous (IV) infusion
Drug: Pembrolizumab — Administered by intravenous (IV) infusion
  Other Names: Keytruda; MK-3475
  Arms: Combination Therapy: Dose Escalation; Combination Therapy: Dose Expansion

SUMMARY:
The purpose of the dose escalation part of the study is to characterize the safety and tolerability of ALN-BCAT as monotherapy and in combination with pembrolizumab; and to determine the recommended dose(s) for expansion (RDFE) of ALN-BCAT as monotherapy and in combination with pembrolizumab. The purpose of the dose expansion part of the of the study is to evaluate the antitumor activity of ALN-BCAT as monotherapy and in combination with pembrolizumab; to characterize the safety and tolerability of ALN-BCAT as monotherapy and in combination with pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Has HCC confirmed histologically or cytologically, or, for patients with liver cirrhosis, clinically by the American Association for the Study of Liver Diseases (AASLD) criteria
* Has had at least one line of systemic therapy for unresectable advanced or metastatic disease
* Has at least one wingless-related integration site (WNT)-pathway activating mutation
* Child-Pugh class A or B7

Exclusion Criteria:

* Has fibrolamellar HCC, sarcomatoid HCC, or mixed cholangio-HCC tumors
* Has symptomatic extrahepatic disease
* Has received anti-cancer therapy or investigational drugs ≤3 weeks prior to the first dose of study drug

Note: other protocol defined inclusion / exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of Adverse Events (AEs) | From the time of first dose of study drug administration to 30-37 days after the last dose
Severity of AEs | From the time of first dose of study drug administration to 30-37 days after the last dose
Dose Escalation: Occurrence of Dose-limiting Toxicities (DLTs) | From the time of first dose of study drug administration up to 21 days
Dose Expansion: Antitumor Activity as assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) | Up to 30-37 Days after the last dose

SECONDARY OUTCOMES:
Concentrations of ALN-BCAT in Plasma | Up to the end of the last study drug administration
  Area Under the Plasma Concentration-time Curve (AUC), Maximum Observed Plasma Concentration (Cmax) Time to Maximum Plasma Concentration (Tmax)
Percent Change in Gene that Encodes ß-catenin Protein (CTNNB1) Messenger Ribonucleic Acid (mRNA) Expression Comparing Pre- treatment with On-treatment Tumor Samples | Up to 30 days
Dose Escalation: Antitumor Activity as assessed by RECIST v1.1 | Up to 30-37 Days after the last dose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals
Locations (21):
- United States (15):
  - Clinical Trial Site, Phoenix, Arizona
  - Clinical Trial Site, La Jolla, California
  - Clinical Trial Site, Los Angeles, California
  - Clinical Trial Site, Jacksonville, Florida
  - Clinical Trial Site, Atlanta, Georgia
  - Clinical Trial Site, Chicago, Illinois
  - Clinical Trial Site, Ann Arbor, Michigan
  - Clinical Trial Site, Rochester, Minnesota
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Cleveland, Ohio
  - Clinical Trial Site, Pittsburgh, Pennsylvania
  - Clinical Trial Site, Dallas, Texas
  - Clinical Trial Site, Houston, Texas
  - Clinical Trial Site, San Antonio, Texas
  - Clinical Trial Site, Richmond, Virginia
- Italy (3):
  - Clinical Trial Site, Milan
  - Clinical Trial Site, Rozzano
  - Clinical Trial Site, Verona
- South Korea (3):
  - Clinical Trial Site, Busan
  - Clinical Trial Site, Seongnam-si
  - Clinical Trial Site, Seoul

IPD SHARING:
Plan to Share IPD: No